CLINICAL TRIAL: NCT05374759
Title: Determination of the Value of Neutrophil Gelatinase-associated Lipocalin and Renal Resistive Index in the Diagnosis and Prognosis of Sepsis-associated Acute Kidney Injury
Brief Title: NGAL and Renal Resistive Index in the Diagnosis and Prognosis of Sepsis-associated AKI
Acronym: NGAL
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ayse Belin Ozer, Prof. Dr., Inonu University
Other Study IDs: AOzer3
Record Dates: First submitted 2022-04-29; First posted 2022-05-16 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Sepsis; Acute Kidney Injury
MeSH Terms: conditions — Sepsis; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients with sepsis who develop AKI
  Interventions: Diagnostic Test: neutrophil gelatinase-associated lipocalin; Diagnostic Test: renal resistive index
- Group 2: Patients with sepsis who do not develop AKI
  Interventions: Diagnostic Test: neutrophil gelatinase-associated lipocalin; Diagnostic Test: renal resistive index

INTERVENTIONS:
Diagnostic Test: neutrophil gelatinase-associated lipocalin — When the patient is diagnosed with sepsis and on the 3rd day of the follow-up, blood samples will be taken and NGAL levels will measured.
Diagnostic Test: renal resistive index — When the patient is diagnosed with sepsis and on the 3rd day of the follow-up, renal resistive index will measure and record.

SUMMARY:
AKI develops frequently in patients hospitalized in the intensive care unit, and the biggest risk factor is sepsis. Creatine, which is traditionally used in the diagnosis of AKI, is affected by many factors, causes the diagnosis to be delayed, and its effect in showing the prognosis is limited. Therefore, there is a need to search for new parameters for early diagnosis and prediction of prognosis. Although many biomarkers studied in blood and urine have been reported in the literature, NGAL has been the most emphasized in terms of both diagnosis and prognosis. Although there are publications on the use of the renal resistive index in the diagnosis in new studies, the place of RRI in the diagnosis has not been determined exactly, and its effect on the prognosis has not been studied. In our study, renal resistive index will be measured by renal ultrasonography at the bedside in patients with sepsis at the time of diagnosis, and NGAL will be studied from the blood of the patients, and their values will be compared in terms of detecting patients with AKI in sepsis and showing prognosis. In summary, if the renal resistive index is superior to serum NGAL and parameters such as creatinine level in showing the diagnosis and prognosis of AKI; Early planning of the patient's treatment with a bedside and non-invasive method will also reduce the cost, considering that ultrasonography is now indispensable for all intensive care units.

DETAILED DESCRIPTION:
In this prospective cross-sectional study, the diagnosis of sepsis (infection+SOFA≥2) and septic shock (lactate>2 in patients with sepsis and vasopressor requirement to keep mean arterial pressure above 65mmHg) were included in our 26-bed mixed intensive care unit, aged 18-70 years. Patients receiving according to sepsis-3 criteria will be included.

Poor abdominal echogenicity, age < 18 years, other conditions causing shock (hypovolemic, cardiogenic, neurogenic), life expectancy shorter than 24 hours, pregnancy, vasospastic disease, intraperitoneal pressure > 15 mm Hg, obstructive renal failure or suspected, presence of arrhythmia , presence of renal artery stenosis, kidney transplant patients, kidney tumor, patients receiving dialysis treatment, single kidney and other kidney abnormalities, presence of coronary artery disease, presence of acute mesenteric ischemia, presence of angiotensin converting enzyme (ACE) inhibition and angiotensin receptor for the last 48 hours Those who use blocking drugs, those with severe acute or chronic renal failure defined as glomerular filtration rate (GFR) < 30 ml/min/1.73m2 will be excluded from the study.

After the patients were diagnosed with sepsis/septic shock, in accordance with the Surviving sepsis 2021 guideline; cultures will be sent and antibiotic, fluid and, if necessary, vasopressor therapy will be started. Standard monitoring of the patients (heart rate, mean arterial pressure, peripheral oxygen saturation, temperature, capillary refill time, perfusion index) will be performed. To determine whether patients develop AKI in the first five days of ICU admission, both creatinine and urine output will be monitored daily according to the KDIGO criteria during the first five days of ICU admission. Patients who developed AKI in our follow-up period after being diagnosed with sepsis/septic shock will be included in Group AKI. Group Control (GK) will be formed from patients who do not develop AKI.

Blood collection for RRI measurement and Serum NGAL level for the study; patients will be diagnosed with sepsis and septic shock, and bundle therapy will be applied for one hour, and after hemodynamic stabilization is achieved (within the first 24 hours). Day 5 RRI measurement and serum NGAL level measurement will be repeated to evaluate the prognosis in patients in group AKI.

The renal resistive index (RRI) will be measured by ultrasound-Doppler. After imaging the kidney in ultrasound mode and checking for renal abnormalities, an arcuate or interlobar artery will be localized and three consecutive Doppler measurements at different points in kidney positions (high, medium, and low) will be performed 3 times in each kidney, resulting in a total of 9 RRI values in each kidney. . The median value of each kidney will be used and the average of the 3 median values of each kidney will be taken.

For serum NGAL level, approximately 10 ml of blood samples taken from the peripheral vein line will be centrifuged at 1500 rpm for 5 minutes and stored at -80 oC.

Patients' age, gender, weight, height, body mass index, concomitant diseases (eg, diabetes mellitus, hypertension, heart failure, COPD, cancer, anemia, intoxications, trauma), source of infection, procalcitonin, c-reactive protein (CRP) ), lactate, circulatory markers, medications (diuretic, vasopressor, inotropic agent, antimicrobial, insulin, colloid, albumin use, blood and blood product transfusion), recent use of contrast media, fluid balance, need for dialysis or hemodiafiltration, mechanical ventilation therapy need, stage of the AKI group according to KDIGO, Acute Physiology and Chronic Health Evaluation (APACHE II) score, Sequential Organ Failure Assesment (SOFA) score, length of hospital stay, renal function before discharge or mortality, and 28-day mortality will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* sepsis
* septic shock

Exclusion Criteria:

* Weak abdominal echogenicity age < 18, other conditions causing shock (hypovolemic, cardiogenic, neurogenic), having a life expectancy of less than 24 hours, pregnancy, vasospastic disease, intraperitoneal pressure > 15 mm Hg, obstructive renal failure or suspected, presence of arrhythmia, presence of renal artery stenosis, kidney transplant patients presence of kidney tumor patients receiving dialysis treatment, solitary kidney and other kidney abnormalities, presence of coronary artery disease, presence of acute mesenteric ischemia, Those who have been using drugs that inhibit angiotensin converting enzyme (ACE) and angiotensin receptor blockers for the last 48 hours, Patients with severe acute or chronic renal failure defined as glomerular filtration rate (GFR) < 30 ml/min/1.73 m2

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with sepsis in ICU.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-12-11 (Actual)

PRIMARY OUTCOMES:
NGAL | at diagnosis
  Blood NGAL
NGAL | at the third days
  Blood NGAL
Renal resistive index | at diagnosis
  renal resistive index guided ultrasound
Renal resistive index | at the third days
  renal resistive index guided ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Ayse Belin B OZER, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Faubel S, Patel NU, Lockhart ME, Cadnapaphornchai MA. Renal relevant radiology: use of ultrasonography in patients with AKI. Clin J Am Soc Nephrol. 2014 Feb;9(2):382-94. doi: 10.2215/CJN.04840513. Epub 2013 Nov 14. PMID 24235286
- [Background] Renberg M, Jonmarker O, Kilhamn N, Rimes-Stigare C, Bell M, Hertzberg D. Renal resistive index is associated with acute kidney injury in COVID-19 patients treated in the intensive care unit. Ultrasound J. 2021 Feb 5;13(1):3. doi: 10.1186/s13089-021-00203-z. PMID 33544258
- [Background] Haitsma Mulier JLG, Rozemeijer S, Rottgering JG, Spoelstra-de Man AME, Elbers PWG, Tuinman PR, de Waard MC, Oudemans-van Straaten HM. Renal resistive index as an early predictor and discriminator of acute kidney injury in critically ill patients; A prospective observational cohort study. PLoS One. 2018 Jun 11;13(6):e0197967. doi: 10.1371/journal.pone.0197967. eCollection 2018. PMID 29889830